CLINICAL TRIAL: NCT01397461
Title: A Phase III 3 Arms, Multicenter, Randomised, Investigator-blind Study to Assess the Efficacy and Safety of Ozenoxacin 1% Cream Applied Twice Daily for 5 Days Versus Placebo in the Treatment of Patients With Impetigo
Brief Title: Efficacy and Safety of Ozenoxacin 1% Cream Versus Placebo in the Treatment of Patients With Impetigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-110880-01
Record Dates: First submitted 2011-07-12; First posted 2011-07-19 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo | interventions — retapamulin; Ointments; ozenoxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ozenoxacin 1% cream (Experimental): 1% cream
  Interventions: Drug: ozenoxacin 1% cream
- ozenoxacin placebo (Placebo Comparator): cream
  Interventions: Drug: ozenoxacin placebo
- retapamulin 1% ointment (Active Comparator): 1% ointment
  Interventions: Drug: retapamulin 1% ointment

INTERVENTIONS:
Drug: ozenoxacin placebo — cream
  Arms: ozenoxacin placebo
Drug: retapamulin 1% ointment — ointment
  Arms: retapamulin 1% ointment
Drug: ozenoxacin 1% cream — 1% cream
  Arms: ozenoxacin 1% cream

SUMMARY:
This is multicenter, randomised, placebo controlled, parallel, blinded (double-blind for ozenoxacin versus placebo comparison and investigator blinded for retapamulin versus placebo comparison), superiority clinical study comparing ozenoxacin cream versus placebo and retapamulin ointment vs placebo, in patients with a clinical diagnosis of non-bullous or bullous impetigo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bullous or non bullous impetigo. The patient has a total affected area comprised between 1-100 cm2 with surrounding erythema not extending more than 2 cm from the edge of any affected area. In case of multiple affected areas the total area will be the sum of each affected area and will not exceed 100 cm2. Additionally for patients < 12 years the total area will not exceed a maximum of 2% of the body surface area.
* Total Skin Infection Rating Scale (SIRS) score of at least 8, including pus/exudate score of at least 1

Exclusion Criteria:

* Has a bacterial infection, which in the opinion of the investigator, could not be appropriately treated by a topical antibiotic.
* Has systemic signs and symptoms of infection (e.g. a fever; defined as an axillary temperature over 37.2 °C (99.0 °F)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (5):
  - Georg Popp, Augsburg
  - Klaus Chelius, Cologne
  - Roland Aschoff, Dresden
  - Diamant Thaci, Frankfurt am Main
  - Stephan Schilling, Mahlow
- South Africa (14):
  - Ismail Mitha, Benoni
  - Johan Lombaard, Bloemfontein
  - Jan Fourie, Dundee
  - Dawie Kruger, George
  - Philip Nel, Hatfield
  - Essack Mitha, Johannesburg
  - J Trokis, Kraaifontein
  - Mohammed Tayob, Middelburg
  - Mashra Gani, Port Elizabeth
  - Zelda Punt, Port Elizabeth
  - Molefe Phayane, Pretoria
  - Gail Todd, Rondebosch
  - Yacoob Vahed, Welkom
  - Christo van Dyk, Worcester

REFERENCES:
- [Derived] Hebert AA, Albareda N, Rosen T, Torrelo A, Grimalt R, Rosenberg N, Zsolt I, Masramon X. Topical Antibacterial Agent for Treatment of Adult and Pediatric Patients With Impetigo: Pooled Analysis of Phase 3 Clinical Trials. J Drugs Dermatol. 2018 Oct 1;17(10):1051-1057. PMID 30365584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 27 sites in the USA, Germany, Romania, Ukraine, and South Africa.
Period: Overall Study
Arm/Group | Ozenoxacin 1% Cream | Ozenoxacin Placebo | Retapamulin 1% Ointment
Started | 155 | 156 | 154
Completed | 153 | 150 | 152
Not Completed | 2 | 6 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was considered the safety populations. The safety population was defined as all patients who had at least one application of study drug.
  One patient was randomised to retapamulin but treated with ozenoxacin. One patient was randomised to retapamulin but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozenoxacin 1% Cream | Ozenoxacin Placebo | Retapamulin 1% Ointment | Total
Number analyzed (Participants) | 156 | 156 | 152 | 464
Age, Customized [Number; unit: Participants]
  2>=years to <12 years | 95 | 94 | 94 | 283
  >=12 years to <18 years | 19 | 18 | 15 | 52
  >=18 years to <65 years | 36 | 40 | 40 | 116
  >=65 | 6 | 4 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 62 | 178
  Male | 100 | 96 | 90 | 286
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 78 | 77 | 78 | 233
  White | 58 | 62 | 50 | 170
  Mixed race | 19 | 15 | 22 | 56
  Asian | 1 | 0 | 2 | 3
  American Indian or Alaska native | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Clinical response (clinical success or clinical failure) at end of therapy (Visit 3) in the intent to treat clinical (ITTC) population.
  Clinical succes at Visit 3 was defined as: SIRS score 0 for exudates/pus, crusting, tissue warmth and pain and no more than 1 each for erythema/inflammation, tissue edema and itching such that no additional antimicrobial therapy in the baseline (Visit 1) affected area is necessary.
  The SIRS is a severity index based on seven signs or symptoms:
  * Exudate/pus
  * Crusting
  * Erythema/inflammation
  * Tissue warmth
  * Tissue oedema
  * Itching
  * Pain
  Each sign/symptom is rated on a scale from 0 to 6:
  0 = absent
  1 2 = mild 3 4 = moderate 5 6 = severe
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Ozenoxacin 1% Cream | Ozenoxacin Placebo | Retapamulin 1% Ointment
Number analyzed (Participants) | 155 | 156 | 154
percentage of participants | 34.8 | 19.2 | 37.7
Statistical Analysis 1: Comparison: Ozenoxacin 1% Cream vs Ozenoxacin Placebo; The treatment comparison was done using only the outcomes of Clinical success and Clinical failure. The p value of the chi square test (without continuity correction) and corresponding 95% asymptotic (Wald) CI for the difference in success rates for the ozenoxacin versus placebo were provided. The analysis was performed to test the superiority of ozenoxacin versus placebo. Text extracted from the statistical analysis plan. No additional data was pre-specified for the statistical comparison; Test type: Superiority or Other; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: AEs were elicited from signing the informed consent to the completion of the clinical study (including the Final Visit) or premature patient withdrawal from the study (10-13 days)
Description: The safety population was defined as all patients who had at least one application of study drug.
  One patient was randomised to retapamulin but treated with ozenoxacin. One patient was randomised to retapamulin but not treated.
Arm/Group | Ozenoxacin 1% Cream | Ozenoxacin Placebo | Retapamulin 1% Ointment
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/156 | 0/152
Other Adverse Events (participants affected / at risk) | 0/156 | 0/156 | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any and all data resulting from the Study will not be presented or published in any form or media by the Institution, Investigator or Research Staff without the prior written consent of Sponsor which consent maybe as directed within the Protocol.